CLINICAL TRIAL: NCT03054415
Title: Anorectal Function and Neuronal-glial-epithelial Unit in Healthy Subjects
Acronym: ANOSAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01541-50
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: neuronal-glial-epithelial unit, anorectal function
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Other)
  Interventions: Procedure: endoscopy

INTERVENTIONS:
Procedure: endoscopy — colonic biopsies during endoscopy and anal manometry with barostat and anal endoflip

SUMMARY:
This study aims to assess the phenotype of the enteric nervous system (enteric neurons) in healthy subjects.

The enteric nervous system (ENS) is composed by enteric neurons and enteric glial cells. There is a cross-talk between ENS and the intestinal epithelial barrier (IEB). ENS and IEB together constitute the neuronal-glial-epithelial unit. This unit has a key role in gut functions. The characteristics and the phenotype of the ENS also change according to age and environmental factors. Similar study is ongoing for patients with Spina Bifida. Anorectal data and phenotype of the neuronal-glial-epithelial unit in healthy subjects is required to assess abnormality of these items in patients with neurological disease including Spina Bifida.

ELIGIBILITY:
Inclusion Criteria:

* subject aged between 18 and 65 years old age and sex matched with the first sixteen patients included and evaluated in the ANOSPIN study
* subject who gave their written consent to participate to the present study
* subject not included in another study
* subject covered by social insurance system

Exclusion Criteria:

* Pregnant or nursing women;
* Anticoagulants therapy or coagulation disorders;
* Past history of anal or rectal surgery
* Crohn disease or ulcerative colitis
* Irritable bowel syndrome according to the Rome III criteria;
* Past history of pelvic radiotherapy
* Pas history of rectal or anal cancer
* Anorectal symptoms : faecal incontinence, constipation, anorectal pain, rectal prolapse;
* CCIS >5 (faecal incontinence);
* Kess Score >9 (constipation);
* Colonic irrigation;
* Use of laxatives;
* Abnormal colonic mucosa
* Period of exclusion;
* Patient under guardianship or unable to give their consent;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2020-02-05 (Estimated)

PRIMARY OUTCOMES:
Number of enteric neurons per ganglion | data collected at the day of endoscopy
  colonic biopsies will be used to study intestinal permeability, colonic inflammation and enteric nervous system

SECONDARY OUTCOMES:
density and activity of the enteric glial cells | data collected at the day of endoscopy
  colonic biopsies will be used to study intestinal permeability, colonic inflammation and enteric nervous system
rectal adaptation | data collected at the day of endoscopy
  rectal adaptation is defined by a volume variation during ascending pressure (phasic distension). It will be performed with a bag connected to electronic barostat
rectal perception | data collected at the day of endoscopy
  It will performed by using 6-point Likert scale ranging from 0 (no sensation) to 6 (intolerable pain)
anal distensiblity | data collected at the day of endoscopy
  It will be performed by using ENDOFLIP
intestinal permeability | data collected at the day of endoscopy
  Biopsy samples collected at the time of colonoscopy will be use within a Ussing Chamber able to assess intestinal permeability. The Ussing chamber is used to measure the short-circuit current as an indicator of net ion transport taking place across an epithelium, such as gut mucosa. The measure will be performed on 2 biopsies from each patient.
macroscopic and microscopic colonic inflammation | data collected at the day of endoscopy
  Colonic inflammation will be assessed during the scope procedure. The physician will assess the normality of the mucosa or not in case of mucosal erythema, ulceration or a decrease of the vascular pattern. Microscopic inflammation will be assessed by the pathologist according to neutrophils infiltration in the gut, crypt abscess, crypt distortion.

CONTACTS AND LOCATIONS:
Overall Officials: Charlène BROCHARD, Md, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Derived] Lefevre C, Le Roy C, Bessard A, Le Berre-Scoul C, Marchix J, Coron E, Le Rhun M, Brochard C, Perrouin-Verbe B, Neunlist M. Region-specific remodeling of the enteric nervous system and enteroendocrine cells in the colon of spinal cord injury patients. Sci Rep. 2023 Oct 6;13(1):16902. doi: 10.1038/s41598-023-44057-y. PMID 37803037
- [Derived] Brochard C, Bouguen G, Olivier R, Durand T, Henno S, Peyronnet B, Pagenault M, Lefevre C, Boudry G, Croyal M, Fautrel A, Esvan M, Ropert A, Dariel A, Siproudhis L, Neunlist M. Altered epithelial barrier functions in the colon of patients with spina bifida. Sci Rep. 2022 May 3;12(1):7196. doi: 10.1038/s41598-022-11289-3. PMID 35505001